CLINICAL TRIAL: NCT05179200
Title: The Effect of Plasma Donation Frequency on Plasma Protein Composition, Inflammation Markers and Psychological Distress - a Randomized Controlled Trial
Brief Title: The Effect of Plasma Donation Frequency on Donor Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 238929
Record Dates: First submitted 2021-12-08; First posted 2022-01-05 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Psychological Distress; Protein Deficiency; Inflammation
Keywords: plasmapheresis; plasma donation; donor health
MeSH Terms: conditions — Protein Deficiency; Inflammation | interventions — Plasmapheresis; Blood Donation

STUDY DESIGN:
Intervention Model Description: Participants/blood donors will be randomized into three donor groups in a 1:1:1 ratio and donate for a 16 week donation period. Group 1 will donate 650 ml plasma (excluding anticoagulant) by plasmapheresis three times every 2 weeks, group 2 will donate 650 ml plasma (excluding anticoagulant) by plasmapheresis once every 14 days and group 3 will donate 450 ml (405-495 ml) whole blood every 3 months.
Who Masked: Outcomes Assessor
Masking Description: The statistical analyses will be blinded with regard to group identity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: "Frequent plasma donors" (Experimental): Donors will donate 650 ml plasma (excluding anticoagulant) by plasmapheresis three times every 2 weeks for 16 weeks.
  Interventions: Procedure: Plasmapheresis
- Group 2: "Regular plasma donors" (Active Comparator): Donors will donate 650 ml plasma (excluding anticoagulant) by plasmapheresis once every 14 days for 16 weeks.
  Interventions: Procedure: Plasmapheresis
- Group 3: "Regular whole blood donors" (Placebo Comparator): Donors will donate 450 ml (405-495 ml) whole blood every 3 months for 16 weeks.
  Interventions: Procedure: Whole blood donation

INTERVENTIONS:
Procedure: Plasmapheresis — Plasma donation
  Other Names: Plasma donation
  Arms: Group 1: "Frequent plasma donors"; Group 2: "Regular plasma donors"
Procedure: Whole blood donation — Blood donation
  Other Names: Blood donation
  Arms: Group 3: "Regular whole blood donors"

SUMMARY:
This project is a randomized controlled non-inferiority study that aims to cover knowledge gaps about the composition and development of plasma proteins, inflammation markers and mental health in Norwegian, voluntary, and unpaid blood donors who donate plasma and blood. We will include 120 male blood donors who are randomized into three groups, the first donating plasma by plasmapheresis 3 times every 2 weeks, the second donating plasma by plasmapheresis every 2 weeks and the third donating whole blood every 3 months. Blood sample analyses are done before, every 2 weeks during the donation period and after the donation period. Questionnaires regarding mental symptoms, Hopkins Symptoms Checklist 25, are done before and after the donation period. The donations extend over 16 weeks and the participants are followed up with blood tests 2 and 4 weeks after the last donation. A plasma sample from each sampling will be stored in an biobank in Innlandet Hospital Trust. The donation frequency are based on the Council of Europe's latest guidelines for plasmapheresis which allow 33 plasma donations per year with at least 96-hour intervals and previous national guidelines. The project is useful to ensure that frequent plasma donations, which are necessary to increase plasma production and the degree of self-sufficiency of plasma products in Norway, do not pose a health risk to blood donors.

The primary objective is to assess the safety of blood donors donating plasma, by comparing the change in total protein and immunoglobulin G concentrations between donors who will be donating plasma 3 times every 2 weeks with donors donating plasma every 2 weeks and blood donors donating regular whole blood every 3 months. The secondary objectives are to compare the concentrations of other plasma proteins and inflammation markers and describe the development of these during plasma and blood donations between the three donations groups, compare the dropout rate and the degree of psychological distress measured by Hopkins Symptoms Checklist 25.

DETAILED DESCRIPTION:
Plasma is the largest single component of blood and makes up about 55% of the total blood volume. It carries the cellular parts of the blood and consists of 90% water, more than 1000 different proteins, and other substances such as minerals, hormones, lipids, and vitamins. The plasma is important for osmotic pressure, intravascular volume, and circulation of hormones, electrolytes, and proteins.

Collected plasma may be used as fresh frozen plasma for transfusion or as plasma for fractionation. Plasma sent for fractionation is further processed into purified therapeutic proteins called plasma-derived medicinal products (PDMPs). Examples of PDMPs are albumin, immunoglobulins, blood coagulation factors like prothrombin complex, and protease inhibitors like α1-antitrypsin. PDMPs are used to treat patients with a wide variety of diseases, for example, congenital diseases like severe combined immunodeficiency, α1-antitrypsin deficiency, or hemophilia. Treatment with PDMPs is often lifelong. Plasma used in transfusion and PDMPs were recently added to the World Health Organization (WHO) Model List of Essential Medicines, underscoring the importance of these products. The demand for plasma and PDMPs is increasing worldwide.

USA is responsible for 70% of the world's source plasma supply. The commercial plasma industry often relies on paid, high-frequency plasma donors, which raises several ethical questions and concerns about donor health. Norway's blood supply is based on voluntary non-remunerated blood donors (VNRBD), which means that a person gives blood, plasma, or cellular components of his/her own free will and receives no payment for it, and this is considered as the safest and most sustainable blood supply.

Current recommendations allow a maximum of 33 plasma donations per year with a minimum 96-hour interval. The collection volume for each plasmapheresis is based on an estimation of the total blood volume calculated according to the International Committee for Standardization in Haematology (ICSH) formula and must never exceed 880 mL plasma. The donation interval is adjusted after measurement of total serum protein (TSP), which is required at the first donation and measured at least annually, as well as serum immunoglobulin G (IgG), which has to be measured at least annually in addition to at every fifth donation. TSP must not be less than 60 g/L, and IgG must not be less than 6.0 g/L. The earlier national guidelines in Norway allowed plasma donations of 650 ml plasma each donation, up to 15 L of plasma every year, and minimum 2 weeks donation interval. At Innlandet Hospital Trust, currently apheresis donors donate every 4 weeks or rarer, and only 324 plasmaphereses were performed in 2019.

The impact of high-frequency plasma donations on plasma protein composition and donor health has not been thoroughly examined. Although high-frequency plasma donation is associated with lower plasma protein levels, donor safety has been ensured by monitoring concentrations of TSP and IgG to adjust donation frequency. A cross-sectional study argued for the safety of long-term intensive donor plasmapheresis of up to 45 l of plasma per year in terms of immunity, red cell and iron metabolism, and cardiovascular risk markers. Another cross-sectional study used pooled plasma samples from different countries with different sampling frequencies and sampling volumes. In this study, however, they found that high-frequency and high-volume plasma donations were associated with a limited ability for plasma proteins, especially immunoglobulins, to return to normal physiological levels. Furthermore, levels of plasma proteins were substantially lower in donors undergoing frequent plasmapheresis than in controls. How these differences in protein concentrations are related to the health of the donors is uncertain.

Hypotheses We hypothesize that high-frequent plasma donation up to every 96 hours is non-inferior compared to plasma donation every 2 weeks and controls regarding donor health measured by the differences in the concentrations of TSP and IgG, and various specific plasma proteins. We also hypothesize that increased levels of inflammation markers and psychological distress are not seen in high-frequency plasma donors compared to plasma donation every 2 weeks and controls.

Study design: Non-inferiority randomized controlled trial of 120 male blood donors who will be randomized to donate plasma with different donation frequency or blood at the Blood Center, Innlandet Hospital Trust; Blood Bank locations include Lillehammer, Hamar, and Elverum over a 16-week intervention period and a 4-week follow-up period. Enrolment of participants will start spring 2022 and donations will start as soon as possible after recruitment.

We have chosen a standard plasma donation volume of 650 ml plasma excluding anticoagulant, which is the maximum plasma donation volume according to the earlier national guidelines. A higher donation volume will increase the possibility to detect a difference in plasma proteins if there is any.

Randomization: Included donors will be randomized into three donor groups in a 1:1:1 ratio. Randomization will be performed as block randomization with a variable block size between 3 and 12.

* Group 1: "Frequent plasma donors". Donors will donate 650 ml plasma (excluding anticoagulant) by plasmapheresis three times every 2 weeks; minimum donation interval is 96 hours.
* Group 2: "Regular plasma donors". Donors will donate 650 ml plasma (excluding anticoagulant) by plasmapheresis once every 14 days.
* Group 3 (control): "Regular whole blood donors". Donors will donate 450 ml (405-495 ml) whole blood every 3 months.

Donors must fulfil criteria for plasma- and blood donations at every donation visit, according to Council of Europe's guideline "Guide to the preparation, use and quality assurance of blood components" and the national "Veileder i transfusjonsmedisin".

Sample size calculation:

The sample size was calculated assuming that before donations TSP (62-78 g/L) and IgG (6.1-14.9 g/L) are within reference intervals. The standard deviations of TSP and IgG in blood donors at Innlandet Hospital Trust are approximately 4 and 2 g/L, respectively. We set the non-inferiority limit for TSP at 2.5 and for IgG at 1.25 g/L. We also assumed a dropout rate of up to 20%. According to these assumptions, we require a sample size of 40 in each donor group (32 participants that can be included in the analyses in each of the study groups). In other words, if there is truly no difference between the standard and experimental treatment, then 32 patients are required per group to be 80% sure that the lower limit of a one-sided 95% confidence interval (or equivalently a 90% two-sided confidence interval) will be above the non-inferiority limit of -2.5 (TSP) or -1.25 (IgG).

Data analysis: Data will be analyzed both on an intent to treat and per-protocol approach. The main outcome of the study will be from the per-protocol analyses where we will include the study participants who complete at least 90% of the scheduled donations. The mean difference between baseline and follow-up of TSP, IgG, other biomarkers, and the scores of the Hopkins symptoms checklist will be compared between the donation groups, using t-tests or other appropriate methods (regression models or ANOVA). In Cox proportional hazards models we will also compare the time until adverse events and/or dropouts between the study groups.

In generalized linear mixed-effects models, we will estimate the interaction between the time (10-time points) of donations and study groups on the concentrations of TSP, IgG, and the other secondary outcomes. In these analyses, we will model the trajectories of the biomarker concentrations between the different study groups. The statistical analyses will be blinded with regard to group identity. We will use Stata and R for these analyses. We will make a detailed plan of analysis before analyzing the main outcomes of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Donors must fulfil criteria for blood- and plasma donation according to Council of Europe's "Guide to the preparation, use and quality assurance of blood components" (14) and "Veileder i transfusjonsmedisin" (16)
2. Age: 18-64 years
3. Sex: Men
4. Estimated blood volume > 4 500 ml
5. Weight >50 kg
6. Donors must have performed at least one plasmapheresis earlier (start at least 2 months after last donation)
7. Good vein quality for plasmapheresis
8. Total serum protein>60 g/L
9. Serum IgG>6.0 g/L
10. Haemoglobin>13.5 g/dL

Exclusion Criteria:

1. Hct >50 %.
2. Medications or medical history not compatible with blood- or plasma donations, for example treatment with angiotensin converting enzyme (ACE) inhibitors, according to guidelines in inclusion criteria

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — We will restrict the participation to male participants to reduce the variability between the study participants. This will increase the statistical power of the study. This also allows higher donation volumes because of higher estimated total blood volume in men (a donation of 650 ml plasma excluding anticoagulant including blood samples, requires an estimated blood volume of minimum 4 500 ml). In subsequent studies, we will include female participants.
Enrollment: 120 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Total serum protein and immunoglobulin G | Measured at week 16 after the donation period
  To compare change from baseline of the TSP (g/L) and IgG (g/L) concentrations at 16 weeks after donations between donors who will be donating plasma 3 times every 2 weeks, donors donating plasma every 2 weeks, and donors who donate whole blood every 3 months.

SECONDARY OUTCOMES:
Other biomarkers | Measured at week 16 after the donation period.
  To compare change from baseline of the concentrations of other biomarkers (reflecting nutritional status, inflammation or other processes related to health and disease, such as plasma proteins, lipids and vitamins) at 16 weeks after donations, and describe the development of these during plasma and blood donations between the three donation groups
Dropout | Week 0-20
  To compare the dropout rate and reasons for dropouts between the three donation groups.
Psychological distress | Measured at week 16 after the donation period.
  To compare the degree of psychological distress, measured by Hopkins Symptoms Checklist 25 before and after donations, between the three donation groups

CONTACTS AND LOCATIONS:
Overall Officials: Tor A Strand, MD/PhD, Principal Investigator — Sykehuset Innlandet HF
Locations (1):
- Innlandet Hospital Trust, Lillehammer, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haugen M, Magnussen K, Aarsland TE, Nissen-Meyer LSH, Strand TA. The effect of donation frequency on donor health in blood donors donating plasma by plasmapheresis: study protocol for a randomized controlled trial. Trials. 2024 Mar 11;25(1):175. doi: 10.1186/s13063-024-08035-7. PMID 38468338
- See also: Full text link — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-024-08035-7
- Available data/document: Study Protocol — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-024-08035-7

DOCUMENTS (2):
  • Statistical Analysis Plan: SOP paper 1 plasma proteins, haematology, AEs and HSCL-25 (2025-02-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT05179200/SAP_000.pdf
  • Statistical Analysis Plan: SOP paper 2 PFAS (2025-09-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT05179200/SAP_001.pdf